CLINICAL TRIAL: NCT02257814
Title: Head Start Classroom-based Approaches and Resources for Emotion and Social Skill Promotion (Head Start CARES)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MDRC (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: HHSP23320072909YC
Record Dates: First submitted 2014-03-25; First posted 2014-10-06 (Estimated); Last update posted 2014-10-06 (Estimated); Status verified 2014-10

CONDITIONS: Teacher Practice; Child Social-Emotional Development

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Control Group (No Intervention): Control group
- Incredible Years (Experimental): incredible years intervention
  Interventions: Behavioral: Incredible Years Teacher Training
- Preschool PATHS (Experimental): Preschool PATHS (Promoting Alternative Thinking Strategies)
  Interventions: Behavioral: Preschool PATHS
- Tools of the Mind (Experimental): Tools of the Mind
  Interventions: Behavioral: Tools of the Mind

INTERVENTIONS:
Behavioral: Incredible Years Teacher Training
  Arms: Incredible Years
Behavioral: Preschool PATHS
  Arms: Preschool PATHS
Behavioral: Tools of the Mind
  Arms: Tools of the Mind

SUMMARY:
The purpose of this study was to deepen the evidence base for interventions that support the social-emotional skills that underlie children's engagement and attention to learning tasks by schools (learning behaviors) and their social interactions with teachers and peers (social behaviors). The study tested three theoretically-distinct approaches to enhancing children's social-emotional development, along with a comprehensive coaching and training model, on a large scale within the Head Start system.

ELIGIBILITY:
Inclusion Criteria:

* Grantees had to have at least 4 centers with a similar racial/ethnic composition
* An equal number of classrooms with full-day or part-day programs
* And a similar mix of four-year-old-only and mixed-age (three-and four-year-old) classrooms.
* Children had to speak English and Spanish.

Exclusion Criteria:

* A grantee was excluded from the sample if it: only ran early Head Start programs
* Only served migrant children
* Was located in a U.S. territory
* Only or mostly provided family child care or home services
* Was more than 100 miles from a "primary airport,"
* Operated fewer than 4 centers with two classrooms each
* Had been in operation for less than 2 years
* Was not in compliance with Head Start Standards
* They were already systematically implementing a social-emotional curriculum or participating in another evaluation study.

Ages: 3 Years to 4 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2670 (Actual)
Dates: Start 2009-04; Primary Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Classroom Climate: Classroom Assessment Scoring System (CLASS) | 0 to 12 months
  Class-level outcome
Teacher Practice: Adapted Teaching Style Rating Scale (TSRS) | 0 to 12 months
  Class-level outcome
Executive Function: Head-to-Toes | 0 to 12 months
  Child-level outcome
Executive Function: Pencil Tap | 0 to 12 months
  Child-level outcome
Social Problem-Solving: Challenging Situations Task | 0 to 12 months
  Child-level outocme
Emotion Knowledge: Emotion Situations and Identification Tasks | 0 to 12 months
  Child-level outcome
Pre-Academic Skills: Academic Rating Scale | 0 to 12 months
  Child-level Outcome
Pre-Academic Skills: Expressive One-Word Picture Vocabulary Test | 0 to 12 months
  Child-level outcome
Pre-Academic Skills: Woodcock-Johnson III | 0 to 12 months
  Child-level outcome
Behavior Regulation: Behavior Problems Index | 0 to 12 months
  Child-level outcome
Social Behaviors: Social Social Skills Rating Scale | 0 to 12 months
  Child-level outcome
Social Behaviors: Cooper-Farran Behavioral Rating Scale- Interpersonal Skills | 0 to 12 months
  Child-level outcome
Learning Behaviors: Cooper-Farran Behavioral Rating Scale- Work-Related Skills | 0 to 12 months
  Child-level outcome

CONTACTS AND LOCATIONS:
Overall Officials: Pamela Morris, Ph.D., Principal Investigator — MDRC/New York University
Locations (1):
- MDRC, New York, New York, United States

REFERENCES:
- [Result] Mattera, S, Lloyd, CM, Fishman, M, and Bangser, M. (2013). A First Look at the Head Start CARES Demonstration: Large-Scale Implementation of Programs to Improve Children's Social-Emotional Competence. OPRE Report 2013-47. Washington, DC: Office of Planning, Research and Evaluation, Administration for Children and Families, U.S. Department of Health and Human Services.